CLINICAL TRIAL: NCT07092410
Title: Surgical or Radiotherapeutic Intervention Concerning Large Singular Stable to Progressive Metastases in Patients With BRAFV600-mutated Melanoma Receiving Treatment With Encorafenib + Binimetinib
Acronym: SuRage-EB
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: SRH Wald-Klinikum Gera GmbH (Other)
Collaborators: Pierre Fabre Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WKG 139175-52; 2024-516073-74-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-07; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Melanoma BRAF V600E/K Mutated
Keywords: BRAFV600-mutated; Melanoma; Encorafenib; Binimetinib; BRAF inhibitor; MEK inhibitor; Braftovi; Mektovi
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to determine PFS (Progression free survival) of individual patients treated with local intervention while continuing therapy with EB.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study. Surgery or radiotherapy or electrochemotherapy in melanoma patients receiving IMP (Other): Local intervention (surgery or radiotherapy or electrochemotherapy) concerning large singular stable to progressive metastases in patients with BRAFV600-mutated melanoma receiving treatment with Encorafenib + Binimetinib
  Interventions: Drug: Encorafenib & Binimetinib Treatment

INTERVENTIONS:
Drug: Encorafenib & Binimetinib Treatment — The SuRage-EB post approval study will evaluate prospectively the potential impact of local treatment of melanoma metastases under encorafenib (E) + binimetinib (B) combination therapy while continuing EB therapy thereafter. It focusses on single melanoma metastases which develop resistance or show no response during EB treatment. These metastases will be treated locally before registration of the patients into the study. Directly after or during local treatment, EB combination therapy will be resumed. Locally treated EB-resistant melanoma cells cannot continue to grow during targeted therapy and the positive response may be prolonged.
  Other Names: Braftovi®; Mektovi®

SUMMARY:
This is an open-label, prospective, single arm study conducted in Germany to investigate local treatment (i.e. surgery or radiotherapy or electrochemotherapy) of metastases showing no response to encorafenib (E) + binimetinib (B) combination therapy and continuation of EB therapy afterwards.

The purpose of this study is to determine PFS of individual patients treated with local intervention while continuing therapy with EB.

DETAILED DESCRIPTION:
The purpose of this prospective study is to evaluate progression free survival (PFS) of patients being treated for a minimum of 3 months with encorafenib and binimetinib and who have non-responding metastases that will be treated with local intervention while continuing combination therapy with encorafenib and binimetinib.

Patients fulfilling the screening-criteria will receive local treatment of 1-3 metastases according to the investigator's decision and according to standard of care. Local treatments are not considered as study related treatments and will be carried out prior to registration. After registration patients will continue approved EB therapy as study treatment.

The aim of the study is to evaluate the effects of local treatment of melanoma metastases that do not respond to EB combination therapy and subsequent continuation of EB therapy on progression-free survival. Local/surgical treatment according to standard of care (= surgery, radiotherapy, electrochemotherapy) will be at the discretion of the investigator. If there are more than one metastasis to be treated locally with different methods authorization of steering committee is required.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all the following criteria:

1. Signed informed consent form
2. Female and male patients ≥ 18 years of age
3. Ability to comply with the study protocol, in the investigator's judgement
4. Ongoing treatment with Encorafenib plus Binimetinib (EB) in accordance with the current Summary of Product Characteristics (SmPC) for a minimum of 3 months
5. ECOG performance status 0-2
6. Life expectancy ≥ 12 weeks
7. Histologically confirmed diagnosis of locally advanced, unresectable or metastatic cutaneous or unknown primary melanoma (inoperable stage III or metastatic stage IV, per AJCC 8 staging)
8. Presence of a BRAFV600-mutation according to a validated test
9. Measurable disease according to RECIST v.1.1, i.e. 1 to 3 locally untreated target lesion(s) to treat with a longest diameter of ≥ 10 mm (lymph node metastases smallest diameter ≥ 15 mm) [TLT; target lesion(s) to treat which are stable or progressive under EB and subject to surgery or electrochemotherapy or radiotherapy within the study] plus ≥ 1 additional target lesion [target lesion(s), which are not subject to surgery or electrochemotherapy or radiotherapy within the study] for continuous measurement Note: Localization of TLTs will be cohortly observed.
10. Availability of RECIST-v1.1-compliant imaging (CT or MRT chest/ abdomen/pelvis and MRT head) within 28 days before initiation of EB treatment outside of the study (= "EB pretreatment") and within 28 days before initiation of surgery or electrochemotherapy or radiotherapy, to assess treatment response under EB pretreatment Note: Steering committee approval is required for older imaging (however, imaging older than 2 months prior to EB initiation is not allowed).
11. Patient must fulfill one of the following conditions (= mixed tumor response) for TLT:

    1. EB in palliative 1st line i. with current response of all metastases according to RECIST v1.1 with exception of 1 to 3 TLT that are stable ii. with current response or stability of all metastases according to RECIST v1.1 with exception of 1 to 3 TLT that are progressing
    2. EB in palliative 2nd line after progression upon checkpoint inhibition in palliative 1st line i. with current response of all metastases according to RECIST v1.1 with the exception of 1 to 3 TLT that are stable ii. with current response or stability of all metastases according to RECIST v1.1 with the exception of 1 to 3 TLT that are progressing

    Notes:
    * Adjuvant BRAFi/MEKi pretreatment with > 6 months of treatment free interval between end of adjuvant and start of palliative 1st line treatment is allowed; any other prior adjuvant therapy is allowed.
    * Inclusion of patients switching from other BRAFi/MEKi to EB within the study treatment line is not allowed.
    * Only for b): BRAFi/MEKi pretreatment in palliative 1st line with direct switch to checkpoint inhibition within this line and without progression is allowed.
    * Mixed tumor response is defined as: some metastases decreasing in size (=responding), some metastases increasing in size (=growing) and/or new metastases appearing, some metastases are stable.
12. TLT must be eligible for treatment with radiotherapy or surgery (R0) or electrochemotherapy; if both, radiotherapy and surgery, required according to national guidelines (e.g., brain metastases) authorization of steering committee is required.
13. Patients must have recovered from all prior treatment related toxicities to NCI CTCAE v5.0 grade ≤ 1, at the time of registration (except for: toxicities not considered a safety risk such as alopecia; stable and non-EB overlapping immune-related (ir) toxicities grade ≤ 2 which are controlled, except ir colitis)
14. Patient with toxicities related to E and/or B [NCI CTCAE v5.0] must have recovered to grade ≤ 1 and be in a stable situation concerning such toxicities
15. Adequate bone marrow, organ function and lab parameters:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    2. Hemoglobin ≥ 9 g/dL without transfusion
    3. Platelet count ≥ 100 x 109/L without transfusion
    4. Creatinine ≤ 1.5 mg/dL, or calculated creatinine clearance (Cockroft-Gault) ≥ 50 mL/min
    5. Serum albumin ≥ 25 g/L
    6. Serum bilirubin ≤ 2.0 x ULN, exception in case of known Gilbert's disease: ≤ 3.0 x ULN
    7. AST/ALT ≤ 2.5 x ULN, exception in case of liver metastases: ≤ 5.0 x ULN
    8. INR/PTT ≤ 1.5 x ULN
16. Adequate cardiac function:

    1. Left ventricular ejection fraction (LVEF) ≥ 50 % as determined by echocardiogram
    2. Triplicate average baseline QTcF interval ≤ 480 msec
17. Negative serum β-hCG test (female patient of childbearing potential only) within 72 hours prior to registration and use of a highly effective contraception for both male and female patients if the risk of conception exists throughout the study and for 4 weeks after study drug discontinuation.

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, should use a highly effective contraception method including:

* Total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation >6 weeks prior to registration; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (>6 months prior to registration); for female patients on the study, the vasectomized male partner must be the sole partner for that patient
* Combination of two of the following:

  1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1 %), for example hormone vaginal ring or transdermal hormone contraception
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  3. Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository

Note:

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to Clinical Trial Facilitation Group guidance. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Exclusion Criteria:

Inclusion Criteria:

Patients may be included in the study only if they meet all the following criteria:

1. Signed informed consent form
2. Female and male patients ≥ 18 years of age
3. Ability to comply with the study protocol, in the investigator's judgement
4. Ongoing treatment with Encorafenib plus Binimetinib (EB) in accordance with the current Summary of Product Characteristics (SmPC) for a minimum of 3 months
5. ECOG performance status 0-2
6. Life expectancy ≥ 12 weeks
7. Histologically confirmed diagnosis of locally advanced, unresectable or metastatic cutaneous or unknown primary melanoma (inoperable stage III or metastatic stage IV, per AJCC 8 staging)
8. Presence of a BRAFV600-mutation according to a validated test
9. Measurable disease according to RECIST v.1.1, i.e. 1 to 3 locally untreated target lesion(s) to treat with a longest diameter of ≥ 10 mm (lymph node metastases smallest diameter ≥ 15 mm) [TLT; target lesion(s) to treat which are stable or progressive under EB and subject to surgery or electrochemotherapy or radiotherapy within the study] plus ≥ 1 additional target lesion [target lesion(s), which are not subject to surgery or electrochemotherapy or radiotherapy within the study] for continuous measurement Note: Localization of TLTs will be cohortly observed.
10. Availability of RECIST-v1.1-compliant imaging (CT or MRT chest/ abdomen/pelvis and MRT head) within 28 days before initiation of EB treatment outside of the study (= "EB pretreatment") and within 28 days before initiation of surgery or electrochemotherapy or radiotherapy, to assess treatment response under EB pretreatment Note: Steering committee approval is required for older imaging (however, imaging older than 2 months prior to EB initiation is not allowed).
11. Patient must fulfill one of the following conditions (= mixed tumor response) for TLT:

    1. EB in palliative 1st line i. with current response of all metastases according to RECIST v1.1 with exception of 1 to 3 TLT that are stable ii. with current response or stability of all metastases according to RECIST v1.1 with exception of 1 to 3 TLT that are progressing
    2. EB in palliative 2nd line after progression upon checkpoint inhibition in palliative 1st line i. with current response of all metastases according to RECIST v1.1 with the exception of 1 to 3 TLT that are stable ii. with current response or stability of all metastases according to RECIST v1.1 with the exception of 1 to 3 TLT that are progressing

    Notes:
    * Adjuvant BRAFi/MEKi pretreatment with > 6 months of treatment free interval between end of adjuvant and start of palliative 1st line treatment is allowed; any other prior adjuvant therapy is allowed.
    * Inclusion of patients switching from other BRAFi/MEKi to EB within the study treatment line is not allowed.
    * Only for b): BRAFi/MEKi pretreatment in palliative 1st line with direct switch to checkpoint inhibition within this line and without progression is allowed.
    * Mixed tumor response is defined as: some metastases decreasing in size (=responding), some metastases increasing in size (=growing) and/or new metastases appearing, some metastases are stable.
12. TLT must be eligible for treatment with radiotherapy or surgery (R0) or electrochemotherapy; if both, radiotherapy and surgery, required according to national guidelines (e.g., brain metastases) authorization of steering committee is required.
13. Patients must have recovered from all prior treatment related toxicities to NCI CTCAE v5.0 grade ≤ 1, at the time of registration (except for: toxicities not considered a safety risk such as alopecia; stable and non-EB overlapping immune-related (ir) toxicities grade ≤ 2 which are controlled, except ir colitis)
14. Patient with toxicities related to E and/or B [NCI CTCAE v5.0] must have recovered to grade ≤ 1 and be in a stable situation concerning such toxicities
15. Adequate bone marrow, organ function and lab parameters:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    2. Hemoglobin ≥ 9 g/dL without transfusion
    3. Platelet count ≥ 100 x 109/L without transfusion
    4. Creatinine ≤ 1.5 mg/dL, or calculated creatinine clearance (Cockroft-Gault) ≥ 50 mL/min
    5. Serum albumin ≥ 25 g/L
    6. Serum bilirubin ≤ 2.0 x ULN, exception in case of known Gilbert's disease: ≤ 3.0 x ULN
    7. AST/ALT ≤ 2.5 x ULN, exception in case of liver metastases: ≤ 5.0 x ULN
    8. INR/PTT ≤ 1.5 x ULN
16. Adequate cardiac function:

    1. Left ventricular ejection fraction (LVEF) ≥ 50 % as determined by echocardiogram
    2. Triplicate average baseline QTcF interval ≤ 480 msec
17. Negative serum β-hCG test (female patient of childbearing potential only) within 72 hours prior to registration and use of a highly effective contraception for both male and female patients if the risk of conception exists throughout the study and for 4 weeks after study drug discontinuation.

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, should use a highly effective contraception method including:

* Total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation >6 weeks prior to registration; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (>6 months prior to registration); for female patients on the study, the vasectomized male partner must be the sole partner for that patient
* Combination of two of the following:

  1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1 %), for example hormone vaginal ring or transdermal hormone contraception
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  3. Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository

Note:

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to Clinical Trial Facilitation Group guidance. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

1. Uveal or mucosal melanoma
2. Presence of untreated brain metastases (exception if this is TLT) Note: Treated brain metastases (stereotactic or surgical intervention) are allowed, if these are stable for > 4 weeks and off corticosteroids for > 3 weeks.
3. Presence of any symptomatic brain and/or leptomeningeal metastases
4. Any previous radiation [including stereotactic radiosurgery (SRS)] therapy involving > 25 % of bone marrow and/or ongoing ≤ 28 days prior to registration (local/surgical intervention excluded)
5. Any major surgery, open biopsy, or significant traumatic injury ≤ 14 days prior to screening Note: Minor surgical procedures should be completed > 7 days prior to registration.
6. Prior treatment with a BRAF- and/or MEK-inhibitor other than EB

   1. in the adjuvant setting and fast relapse (i.e., treatment free interval between adjuvant and palliative 1st line ≤ 6 months) is not allowed
   2. in the palliative setting is not allowed Exception: Pretreatment with BRAF- plus MEK-inhibition in palliative 1st line and direct switch to checkpoint-inhibition within this line without progression
7. Any prior systemic chemotherapy for the current melanoma disease Note: Chemotherapy given as part of isolated limb perfusion, regional or intralesional treatment will not be considered systemic treatment
8. Any use of an investigational agent ≤ 28 days or ≤ 5 half-lives (minimum 14 days) or an approved medication except of E + B prior to registration, whichever is shorter
9. Any intake of the following foods/supplements within ≤ 7 days prior to registration:

   1. St. John's wort or hyperforin
   2. Grapefruit and Grapefruit juice
10. Any condition that would interfere with the planned radiotherapy or surgery or electrochemotherapy of TLT Note: If one of these therapies is without interference this should be performed in the study.
11. Any contraindication against the radiotherapy or surgery or electrochemotherapy of TLT Note: If one of these therapies is without contraindication this should be performed in the study.
12. Known hypersensitivity to any components of the study treatment
13. Any malabsorption condition that would alter the absorption of orally administered medications
14. Inability to swallow oral medication
15. History of allogeneic bone marrow or organ transplant requiring use of immunosuppressive medication
16. Known positive serology for HBV, HCV and/or HIV
17. Any active infection requiring systemic antibiotic therapy ≤ 2 weeks prior to registration
18. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma with intraocular pressures > 21 mm HG or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
19. Impaired cardiovascular function or clinically significant cardio-vascular diseases, including the following:

    1. Myocardial infarction ≤ 6 months prior to registration
    2. Severe/unstable angina pectoris ≤ 6 months prior to registration
    3. Cerebrovascular accident or transient ischemic attack ≤ 6 months prior to registration
    4. History of symptomatic congestive heart failure (NYHA stage ≥ 2)
    5. History of congenital long QT syndrome or mean QTcF > 480 msec or uncorrectable electrolyte abnormalities
    6. Uncontrolled arterial hypertension despite medical treatment (patients with a history of hypertension controlled to ≤ grade 1 with anti-hypertensives are eligible)
    7. Uncontrolled or clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree atrioventricular [AV] block without a pacemaker)
20. Neuromuscular disorders that are associated with elevated creatine phosphokinase (CK) (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
21. Previous or concurrent malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell skin cancers (adequate wound healing prior to registration)
    2. in situ carcinoma of the cervix, treated curatively and without evidence of recurrence for at least 3 years prior to registration
    3. or other solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to registration
22. Known alcohol or drug abuse
23. Any medical, psychiatric, cognitive or other conditions that would, in the investigator's judgement, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results
24. Participation in another trial (non-interventional studies are allowed) within 30 days prior to screening
25. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive β-hCG laboratory test
26. Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) after local treatment (radiotherapy / surgery / electrochemotherapy) | From enrollment up to end of treatment period after 52 weeks maximum.
  The purpose of this study is to determine PFS of individual patients treated with local intervention while continuing therapy with EB.

SECONDARY OUTCOMES:
Overall Response Rate (ORR), Disease Control Rate (DCR), Duration of Response (DoR), Duration of Disease Control (DoDC), Duration of Stable Disease (DoSD) | From enrollment up to end of treatment period after 52 weeks maximum.
progression-free survival rate (PFSR) at 1 year after local treatment (radiotherapy / surgery /electrochemotherapy) | From enrollment up to end of treatment period after 52 weeks maximum.
time to treatment failure (TTF) | From enrollment up to end of treatment period after 52 weeks maximum.
overall survival (OS) | From enrollment up to end of treatment period after 52 weeks maximum.
Quality of Life (QoL) | From enrollment up to end of treatment period after 52 weeks maximum.
  Quality of Life (QoL) by means of questionnaires FACT-M, EQ-5D-5L, EORTC QLQ-C30
safety / toxicity according to CTCAE Version 5.0 criteria | From enrollment up to end of treatment period after 52 weeks maximum.
  safety / toxicity according to CTCAE Version 5.0 criteria:
  * (Serious) Adverse events (overall and differentiated by patients undergoing surgery, radiotherapy or electrochemotherapy)
  * Adverse reactions concerning surgery, radiotherapy, electrochemotherapy, encorafenib and binimetinib

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaatz, PD Dr. med. habil., Study Director — SRH Wald-Klinikum Gera GmbH

IPD SHARING:
Plan to Share IPD: Yes